CLINICAL TRIAL: NCT01972633
Title: Endovenous Treatment of the Saphenous Vein With Biolitec 1470nm Laser Versus Vnus Closure Fast
Brief Title: Endoluminale Obliteration Der Stammvene Mit Dem 1470nm Laser Versus VNUS Closure Fast
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig Boltzmann Institute for Operative Laparoscopy (Other)
Responsible Party: Principal Investigator, Dr. Markus Schreiner, Oberarzt, Ludwig Boltzmann Institute for Operative Laparoscopy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Boltzmann-001
Record Dates: First submitted 2012-12-04; First posted 2013-10-30 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Venous Insufficiency
Keywords: endovenous treatment; Laser, Vnus Closure Fast; Varicosis; great saphenous vein; small saphenous vein; Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1470nm Laser (Active Comparator): Patient with varicose vein treated with 1470nm Laser (Biolitec)
  Interventions: Procedure: Laser; Procedure: Radiofrequency
- VNUS Closure Fast (Active Comparator): Patient with varicose vein treated with VNUS Closure Fast (Radiofrequency System)
  Interventions: Procedure: Laser; Procedure: Radiofrequency

INTERVENTIONS:
Procedure: Laser — Endovenous Laser (1470nm) ablation of great or small saphenous vein
Procedure: Radiofrequency — Endovenous Radiofrequency (VNUS Closure Fast) of great or small saphenous vein

SUMMARY:
There is a difference concerning obliteration rate and postoperative pain after treatment of the saphenous vein with 1470nm laser or VNUS Closure Fast (=radiofrequency method) .

DETAILED DESCRIPTION:
The endovenous treatment of the insufficient saphenous vein (large saphenous vein and small saphenous vein) is a standard procedure for years. There are different methods that cause an obliteration of the vein using heat. The adventage of these methods are low rates of minor and major complications compared to classic open surgery. There are also advantages concerning cosmetic and recurrence of varicous veins. Actually there are two different methods for the endovenous obliteration of the saphenous vein - lasers with wavelength of 1470nm or 1320nm and the radiofrequency method. The objective of this study is to compare these two different methods concerning postoperative pain, obliteration rate and the rate of pleased patients in 140 patients. All patients get an venous ultrasound investigation to determine the stadium of venous insufficiency. There are consecutive ultrasound investigations 10 days, 3 months and 12 months after surgical treatment.

In this study there are no additional risk factors for the included study patients except the risk of surgery.

ELIGIBILITY:
Inclusion Criteria:

* varicosis of great saphenous vein Hach-classification II-III (CEAP-classification: C3-4EPAS2-3PR and/or varicosis of small saphenous vein der Hach-classification I-III CEAP-classification: C3-4EPAS4PR)
* maximum diameter of the great saphenous vein of 15mm maximum diameter of the small saphenous vein of 12mm

Exclusion Criteria:

* surgical treatment of the saphenous vein in the past
* sclerotherapy of the saphenous vein in the past
* phlebitis or thrombosis of the saphenous vein
* surgical treatment of an venous ulcer in the past
* postthrombotic syndrome
* erysipelas of the leg in the past
* chronic treatment with pain-killers or chronic alcoholism
* pregnancy
* drug allergy against painkillers that are used in this study
* spinal anesthesia not possible
* compression bandage not possible
* patients with polyneuropathy
* patients with chronic pain
* persons that do have a connection or persons that are working for one of the jused companies (Laser or VNUS Closure Fast)
* participation on an other clinical trial that can interfere with this clinical trial
* missing written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Pain | day 0
  Pain (visual analogue scale) on the day of treatment

SECONDARY OUTCOMES:
Obliteration of the treated vein (GSV or SSV) | day 10, month 3, month 12
  An ultrasound investigation of he treated vein is done to find out if the treated vein is fully obliterated or not. If it is not fully obliterated we want to find out if there is any pathological reflux in the vein.
Patient´s satisfaction after the intervention | day 10, month 3, month 12
  The patient is asked about his/her satisfaction after intervention. This is measured on a numeric scale from 1 to 5 (like schoolmarks in austria or germany). 1=very good, 2=good, 3=average, 4=not so good, 5=bad)

OTHER OUTCOMES:
paresthesia of the lower leg after intervention | day 10, month 3, month 12
  patients are asked if there is any paresthesia of the lower leg - "yes" or "no"

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schreiner, Principal Investigator — 2.Chirurgische Abteilung AKh Linz GesmbH; Andreas Shamiyeh, Study Chair — 2. Chirurgische Abteilung AKh Linz GesmbH
Locations (1):
- 2.Chirurgische Abteilung AKh Linz GesmbH, Linz, Upper Austria, Austria